CLINICAL TRIAL: NCT00020644
Title: Phase I Study of Continuous Infusion Gemcitabine
Brief Title: Continuous Infusion Gemcitabine in Treating Patients With Advanced Metastatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advocate Lutheran General Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: LGH-3000; CDR0000068691 (Registry Identifier: PDQ (Physician Data Query)); NCI-V01-1660
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2004-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of gemcitabine given as a continuous infusion in treating patients who have advanced metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of continuous infusion gemcitabine in patients with metastatic malignancies.
* Determine the toxicity profile of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients on dose levels 1-5 receive gemcitabine IV continuously over 72 hours on week 1. Patients on dose levels 6 and 7 receive gemcitabine IV continuously over 72 hours on weeks 1-3. Courses repeat every 2 weeks (for patients on dose levels 1-5) and every 4 weeks (for patients on dose levels 6 and 7) in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of an advanced metastatic malignancy for which no curative therapy exists

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Pulmonary:

* Corrected DLCO at least 60% expected

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior short-infusion gemcitabine allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Brian L. Samuels, MD, Study Chair — Advocate Lutheran General Hospital
Locations (1):
- Lutheran General Cancer Care Center, Park Ridge, Illinois, United States